CLINICAL TRIAL: NCT04864184
Title: The Effects of Different Breathing Styles on Post High-Fat Meal Blood Vessel Function
Brief Title: Effects of Breathing Patterns on Post-prandial Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7374
Record Dates: First submitted 2021-03-29; First posted 2021-04-28 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: Breathing; Yogic breathing
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Each participant will complete 2 different sessions in random order.
Masking Description: Participants will be blinded to the respiratory rates being practiced during each study visit. Breathing patterns will be completed in random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing intervention (Experimental): Participants will complete 2-minute breathing exercises following the Breathing App every 15 minutes during a 4-hour postprandial period following high-fat meal consumption.
  Interventions: Behavioral: Normal physiologic rate breathing; Behavioral: Slow breathing

INTERVENTIONS:
Behavioral: Normal physiologic rate breathing — 2-minute breathing exercises will be completed every 15 minutes.
Behavioral: Slow breathing — 2-minute breathing exercises will be completed every 15 minutes.

SUMMARY:
The purpose of this study is investigate the effects of two different breathing styles on postprandial vascular function and oxidative stress markers. Participants will complete 2 breathing conditions in random order.

ELIGIBILITY:
Inclusion Criteria:

• Male participants ages 18-35 years

Exclusion Criteria:

* Infection within the previous 4 weeks
* Renal disorders
* Any cardiovascular disorders such as prior myocardial infarction, known coronary artery disease, personal history of stroke, heart failure, cardiac arrhythmias
* Chronic obstructive pulmonary disease
* Diabetes
* Inflammatory bowel disease
* HIV, rheumatoid arthritis, chronic or other inflammatory conditions
* Currently taking steroids or other anti-inflammatory medications
* Current use of nonsteroidal anti-inflammatory drugs
* Smoking
* Stage 2 hypertension or higher (systolic BP of 140 mm Hg or higher and/or diastolic BP of 90 mm Hg or higher)
* Lactose intolerance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilation | At baseline and at again 1, 2, 4 hours post high-fat meal consumption
  Ultrasound-derived images of the brachial artery pre- and post-suprasystolic cuff inflation will yield flow-mediated dilation values. These are indices are endothelium-dependent vasodilation.
Changes in oxidative stress | Once at baseline and again at 1, 2, and 4 hours post high-fat meal consumption.
  Blood draws will be performed and samples will be processed and stored for future biochemical analysis of blood markers indicative of oxidative stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Physiology Laboratory-Texas State University, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hunter SD, Bernardi L, McAllister MJ, John D, Rahimi M, Lopez MR. Device-guided slow breathing alters postprandial oxidative stress in young adult males: A randomized sham-controlled crossover trial. Nutr Metab Cardiovasc Dis. 2023 Jan;33(1):203-209. doi: 10.1016/j.numecd.2022.10.002. Epub 2022 Oct 10. PMID 36344308